CLINICAL TRIAL: NCT05657106
Title: Kentucky Outreach Service Kiosk (KyOSK): Reducing HIV, HCV, and Overdose Risk in Rural Appalachia Through Harm Reduction Kiosks
Brief Title: Kentucky Outreach Service Kiosk (KyOSK): Reducing HIV, HCV, and Overdose Risk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: April M Young (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, April M Young, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KyOSK; 1R01DA055872 (NIH)
Record Dates: First submitted 2022-11-03; First posted 2022-12-20 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Opioid-Related Disorders; Hepatitis C (HCV); Human Immunodeficiency Virus (HIV); Drug Overdose; Substance Abuse; Intravenous Drug Usage; Opiate Substitution Treatment; Sexually Transmitted Diseases
MeSH Terms: conditions — Opioid-Related Disorders; Hepatitis C; Acquired Immunodeficiency Syndrome; Drug Overdose; Substance-Related Disorders; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Type 1 hybrid effectiveness study involving a community-level, controlled quasi-experimental trial and a mixed methods evaluation of implementation outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Syringe Service Program Plus a Harm Reduction Kiosk Intervention (Experimental): The intervention to be implemented in the intervention county involves enhancing its existing SSP model with a KyOSK. The intervention county SSP operates identically to the comparison county. As in the comparison county, a card reader will be installed in the intervention county SSP at the beginning of the study to provide objective data on visits and supply access. The KyOSK will resemble a vending machine. The KyOSK will include harm reduction, wound care, hygiene, and other supplies; offer overdose education and other content; a sharps container with a device to obtain data on syringe disposal; and an innovative call-back feature for care navigation by recovery coaches. While the KyOSK is operating, the intervention county will operate its traditional SSP 40 hours/week.
  Interventions: Behavioral: Harm reduction kiosk
- Syringe Service Program (No Intervention): The comparison county SSP operates in the local health department and provides syringes, cookers/cottons, naloxone, wound care kits, condoms and lubricant, snacks, drinks, and sharps containers. A peer support specialist is present for consultation with clients upon request during SSP hours. The SSP will expand it hours from 3 hours/week to 40 hours/week at the same time the intervention county receives its KyOSK, to be comparable. SSP clients who enroll in the study will receive a swipe card linked to their SSP client identification. Card readers will be installed in the SSP for clients to swipe upon entry. Staff will provide clients with the same menu of supplies as those in the KyOSK and the same supply/time interval limits will be imposed. SSP clients will receive a resource guide.

INTERVENTIONS:
Behavioral: Harm reduction kiosk — The intervention involves enhancing an existing staffed harm reduction program (syringe service program) located in a local health department with a Kentucky Outreach Service Kiosk (KyOSK).
  Arms: Syringe Service Program Plus a Harm Reduction Kiosk Intervention

SUMMARY:
This study will test the effectiveness, implementation outcomes, and cost effectiveness of a community-tailored, harm reduction kiosk in reducing HIV, hepatitis C, and overdose risk behavior in rural Appalachia. The proposed project will take place in two counties in Appalachian Kentucky, an epicenter for the intertwined national crises of injection drug use, overdoses, and hepatitis C.

DETAILED DESCRIPTION:
This is a Type 1 hybrid effectiveness study involving a community-level, controlled quasi-experimental trial to assess the impact of a community-tailored harm reduction kiosk on HIV, HCV, and overdose risk in rural Appalachia, and a mixed methods evaluation of implementation outcomes. The trial will compare the standard local syringe service program (SSP) design (brick-and-mortar, staffed by department of health staff) to an enhanced model involving a harm reduction kiosk + standard SSP. The kiosk, referred to as the KyOSK (Kentucky Outreach Service Kiosk) will be tailored through a community-engaged adaptation process. For evaluation of the KyOSK's impact on HCV and overdose risk behavior, the investigators will enroll 750 People Who Use Drugs (PWUD) in the intervention (n=425) and comparison (n=325) counties, collectively referred to as the kiosk trial cohort. The kiosk trial cohort will be recruited from three sources: existing cohorts of PWUD, SSPs, and peer-referral. Throughout the trial and following the implementation outcome framework (IOF) measurement model by Proctor et al., acceptability, appropriateness, fidelity, cost, penetration, and sustainability will be assessed using a combination of validated scales, qualitative interviews, checklists, invoices, and program data. Following the trial, the investigators will use data collected from the kiosk cohort and implementation outcome assessment (primarily cost and reach) in a dynamic, deterministic model of HCV transmission and overdose to examine the impact and cost-effectiveness of the KyOSK model.

ELIGIBILITY:
Inclusion Criteria:

Individuals are eligible if they are:

* age 18 or older,
* live in the intervention or comparison county, and
* have engaged in injection or non-injection illicit drug use to get high in the past 6 months (excluding marijuana, alcohol, and tobacco).

Exclusion Criteria:

Individuals are not eligible if they meet any of the exclusion criteria:

* being under the age of 18,
* not living in the intervention or comparison county,
* having not engaged in injection or non-injection illicit drug use to get high in the past 6 months (excluding marijuana, alcohol, and tobacco),
* not being able to speak or understand English,
* conviction in the past 10 years of a violent crime (i.e., murder, manslaughter, rape, robbery, and /or aggravated assault) or stalking,
* current charges of violent crime or stalking, or
* having plans to move out of the study counties in the next 6 months, or residing in an inpatient facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in syringe coverage for injections | Measured at baseline and then every 6 months up to 5 years
  Self-reported number of injections in the past 30 days where a clean syringe was used divided by the total number of injections in the past 30 days
Change in harm reduction program supplied syringe coverage for injections | Measured at baseline and then every 6 months up to 5 years
  Number of syringes obtained at the SSP and/or KyOSK in the past 30 days (obtained from card swipe/supply dispensing data)
Change in SSP / KyOSK-provided syringe coverage for injections | Measured at baseline and then every 6 months up to 5 years
  Self-reported number of injections in the past 30 days where a clean syringe from the [KyOSK/SSP] was used divided by the total number of injections in the past 30 days

SECONDARY OUTCOMES:
Change in frequency of receptive syringe sharing among participants who inject drugs | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) frequency of using a syringe that had been previously used by someone else (continuous; number and proportion)
Change in frequency of distributive syringe sharing among participants who inject drugs | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) frequency of providing a used syringe to someone else (continuous)
Change in number of people with whom person shared syringes and injection equipment | Measured at baseline and then every 6 months up to 5 years
  Self-reported number of people participant shared syringes and other injection equipment with in the past 30 days (continuous)
Change in frequency of syringe reuse among participants who inject drugs | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) number of times re-using syringes (continuous)
Change in frequency of safe syringe disposal among participants who inject drugs | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) disposal of syringes in a sharps container or syringe exchange program (binary)
Change in frequency of condom-less anal and/or vaginal sex | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) frequency of anal or vaginal sex without a condom (continuous; number and proportion of all sex events)
Change in frequency of overdose | Measured at baseline and then every 6 months up to 5 years
  Self-reported number of times overdosed in the past 6 months (continuous).
Change in use of naloxone during overdose events by participants who witnessed an overdose | Measured at baseline and then every 6 months up to 5 years
  Self-reported number of times overdosed in the past 6 months (continuous)
Change in number of days carrying naloxone | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) frequency of carrying naloxone (continuous)
Change in number of times contacting or visiting a pharmacy to obtain naloxone | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 6 months) frequency of naloxone seeking at a pharmacy (continuous)
Change in number of days on medications for opioid use disorder (MOUD) among participants who use opioids to get high | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) frequency of being on MOUD (continuous)
Change in frequency of use of harm reduction services among participants who inject drugs | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) frequency of providing a used syringe to someone else (continuous, number and proportion of syringes)
Change in frequency of use of fentanyl test strips among participants who use drugs | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) frequency of using a fentanyl test strips (binary)
Change in frequency of engagement in overdose protective behaviors among participants who use drugs | Measured at baseline and then every 6 months up to 5 years
  Self-reported recent (past 30-day) frequency of engaging in overdose protective behaviors

CONTACTS AND LOCATIONS:
Overall Officials: April M Young, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young AM, Jahangir T, Westneat S, Cheatom C, Fallin-Bennett A, Fanucchi LC, Freeman PR, Havens JR, Knudsen HK, McCollister KE, Stitzer S, Stone J, Vickerman P, Livingston MD. Preferences for harm reduction vending machine design among rural people who use drugs. Drug Alcohol Depend Rep. 2025 Oct 31;17:100391. doi: 10.1016/j.dadr.2025.100391. eCollection 2025 Dec. PMID 41322680
- [Derived] Young AM, Havens JR, Cooper HLF, Fallin-Bennett A, Fanucchi L, Freeman PR, Knudsen H, Livingston MD, McCollister KE, Stone J, Vickerman P, Freeman E, Jahangir T, Larimore E, White CR, Cheatom C, Community Staff K, Design Team K. Kentucky Outreach Service Kiosk (KyOSK) Study protocol: a community-level, controlled quasi-experimental, type 1 hybrid effectiveness study to assess implementation, effectiveness and cost-effectiveness of a community-tailored harm reduction kiosk on HIV, HCV and overdose risk in rural Appalachia. BMJ Open. 2024 Mar 1;14(3):e083983. doi: 10.1136/bmjopen-2024-083983. PMID 38431295